CLINICAL TRIAL: NCT03463148
Title: Validation of a Sensor for Non-Invasive Measurement of Vital Signs, Hemodynamic Parameters and Time-Dependent Physiological Waveforms
Brief Title: Validation of a Sensor for Non-Invasive Measurements
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TS-IRB-0003
Record Dates: First submitted 2018-01-31; First posted 2018-03-13 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: CHF; Renal Disease; Hypertension
MeSH Terms: conditions — Kidney Diseases; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- 1: Men/Women who meet the inclusion/exclusion criteria of this protocol.

SUMMARY:
Subjects will be measured with both a sensor and a reference device

DETAILED DESCRIPTION:
Subjects will participate in a study measuring a single set of paired values. In this case, measurements will take roughly 2-30 minutes to complete, and will involve: 1) attaching the sensor on the subject; 2) attaching one or more reference devices to the subject; 3) making measurements with both the sensor and reference device, either simultaneously or sequentially; and 4) collecting and analyzing the paired value.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 (eighteen) years of age at screening.
2. Subject and/or legally authorized person/representative is willing to undergo the Informed Consent process prior to enrollment in the study.
3. Subject selection will not be based on age, height, or weight.
4. Subject is a candidate for this study based on the PI's opinion and knowledge of the subject's condition as well as the features of the investigational device tested during the study.

Exclusion Criteria:

1. Subject is participating in another clinical study that may affect the results of either study.
2. Subjects that are pregnant will not be included in the study.
3. Subject is unable or not willing to wear electrode patches as required for a period of up to 168 hours.
4. Subject is considered by the Principal Investigator to be medically unsuitable for study participation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Men and women over 22 years of age
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Comparison of Blood Pressure Measurement from Sensor with Human Auscultation measurement of Blood Pressure. | 3-36 Months
  Comparison of Blood Pressure Measurement from Sensor with Human Auscultation measurement of Blood Pressure. Specifically, Systolic Blood Pressure and Diastolic Blood Pressure with units of millimeters of mercury (mmHg) will be compared.
Fluids | 3-36 Months
  Observation of fluid measurement from Sensor (ohms)
Heart Rate | 3-36 Months
  Observation of heart rate measurement from Sensor (beats/min)
Heart Rate Variability | 3-36 Months
  Observation of heart rate variability from Sensor (milliseconds)
Respiration Rate | 3-36 Months
  Observation of respiration rate from Sensor (breaths/min)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Banet, PhD, Principal Investigator — Baxter Healthcare Corporation
Locations (1):
- toSense, Inc. Headquarters, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No